CLINICAL TRIAL: NCT05324488
Title: Diabetes Registry Graz for Biomarker Research
Acronym: GIRO
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: HS-2015-01
Record Dates: First submitted 2021-09-29; First posted 2022-04-12 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Type1diabetes; Type 2 Diabetes; Adiposity
Keywords: cohort study
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples Without DNA — Urinary, plasma and serum samples are collected for future analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Type 1 Diabetes: Patients with diagnosed type 1 diabetes mellitus
  Interventions: Other: No intervention
- Type 2 Diabetes: Patients with diagnosed type 2 diabetes mellitus
  Interventions: Other: No intervention
- Adipositas: Obese patients with a BMI > 30kg/m2
  Interventions: Other: No intervention
- Lipid metabolism disorder: Patients with disorder of lipid metabolism
  Interventions: Other: No intervention
- Type 3 Diabetes Mellitus: Patients with diagnosed type 3 diabetes mellitus
  Interventions: Other: No intervention
- Maturity onset diabetes of the young (MODY): Patients with diagnosed MODY
  Interventions: Other: No intervention
- Late onset diabetes of the adult (LADA): Patients with diagnosed LADA
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — In this registry no intervention is carried out

SUMMARY:
The Diabetes registry for biomarker research Graz is a prospective cohort-study including subjects with type 1 and type 2 diabetes, rare types of diabetes, obesity and dyslipidemia, aiming to collect data, blood and urine samples of all subjects on an annual basis.

DETAILED DESCRIPTION:
Obesity and diabetes represent probably the most challenging threat to public health in the 21st century.

Despite well-controlled established cardiovascular risk factors, the residual risk in subjects with diabetes mellitus is significantly higher than the risk in those without the condition and it is well established that current risk prediction models for cardiovascular disease using established risk factors do not fully explain the future cardiovascular risk.

Therefore, biomarker for better risk stratification are needed, in particular in subjects with diabetes mellitus. Prospective cohorts, meticulously clinically phenotyping subjects, regularly following them and collecting biomarker samples is one key approach for finding new biomarker panels, that are predictive of treatment response and future micro- and macrovascular complications.

The Diabetes registry for Biomarker Research Graz was initiated in November 2015. Subjects with type 1 and type 2 diabetes, rare types of diabetes, obesity or dyslipidemia are recruited in the outpatient clinic for Diabetes, Lipid and Metabolic Disorders at the University Clinic Graz or in the Rehabilitation Center St. Radegund.

As of September 2021, 1250 subjects are recruited. Blood and urine samples samples are collected at baseline and at annual follow up visits as well as data on medical history, diagnoses and medication.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 99 years
* Informed consent has to be given in written form
* At least one of the following diseases:
* Type 1 diabetes
* Type 2 diabetes
* Type 3 diabetes
* Maturity onset diabetes of young (MODY)
* Late onset diabetes of the adult (LADA)
* Adipositas (BMI > 30kg/m2)
* Lipid metabolism disorder

Exclusion Criteria:

* No written informed consent
* No willingness to participate in this registry

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with different types of diabetes as well as obesity and lipid metabolism disorder are observed in this registry.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-10-21 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-02-01 (Estimated)

PRIMARY OUTCOMES:
Biomarker identification | Over entire period of registry (20 years)
  Identification of biomarker panels that allow prediction of future micro- and macrovascular disease and events.
  Changes of these biomarkers over time in a selected, defined cohort will be reported.

SECONDARY OUTCOMES:
Biomarker validation | Over entire period of registry (20 years)
  Validation of suggested biomarkers in the field of diabetes complications.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sourij, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No